CLINICAL TRIAL: NCT05993208
Title: Correlation Between Optical Coherence Tomography and Multifocal Electroretinogram Findings With Visual Acuity After Vitrectomy Surgery for Retinal Detachment
Brief Title: Correlation Between OCT and mFERG Findings With VA After Vitrectomy Surgery for Retinal Detachment
Status: Completed | Type: Observational
Sponsor: New Valley University (Other)
Collaborators: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Kamel Ahmed Hassan, lecture, New Valley University
Other Study IDs: CBOCT&MFERG&VA-VRD
Record Dates: First submitted 2023-07-28; First posted 2023-08-15 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-08

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: optical coherence tomography,multifocal electroretinogram. VA measurment — retinal photography

SUMMARY:
Correlation between optical coherence tomography and multifocal electroretinogram findings with visual acuity after vitrectomy surgery for Retinal detachment.

DETAILED DESCRIPTION:
Although the anatomical success rate of vitreoretinal surgery has improved over the last decade, visual results remain compromised? Patients with macula-off retinal detachments (RDs) can have poor visual recovery, specific color vision defects, or metamorphopsia postoperatively despite successful retinal reattachment. In these cases, subtle changes in the foveal structure may be causing visual disturbances that can be difficult to identify during standard clinical examinations such as slit lamp biomicroscopy or binocular indirect ophthalmoscopy .reported a possible association between incomplete visual recovery and the presence of residual subretinal fluid (SRF) postoperatively.

Optical coherence tomography (OCT) is a non-invasive technique that provides information about the morphology of the retina, and especially of the macular area in vivo. Some studies support the idea that OCT determines structural changes in the macula that are correlated with subjective visual function, including visual acuity (VA) in patients with vitrectomy for retinal detachment. Additionally, multifocal electroretinogram (m fERG) evaluation can be helpful in assessing macular function in post-vitrectomy. However, to date, there are relatively few reports concerning the combined use of OCT and m fERG for the correlation between retinal morphology and function of the macula in patients with vitrectomy for retinal detachment surgery. The purpose of our study is to determine whether a significant correlation exists between the amplitude of m fERG, visual acuity, and the morphological OCT changes by in the macula after vitrectomy for retinal detachment

ELIGIBILITY:
Inclusion Criteria:

* patients with successful vitrectomy for retinal detachment.

Exclusion Criteria:

* The patients who had vitrectomy for reasons other than retinal detachment surgery
* Patients who had done scleral buckle surgery
* Patients with media opacity are prevented from doing retina imaging.
* Failed or recurrent vitrectomy surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective observation (analytic) study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
CMT,BCVAand mf-ERG were recoreded in 40 eyes of 40 patintes with vitrectomy for retinal detchament surgery . | 6 months
  Each 10 um increase in central (CMT) associated by how increase decimal in Best corrected visual acuity and by how nV/deg2 increase multifocal electroretinogram in these eyes .
BCVA(best corrected visual acuity) | 6 Month
  Best corrected Visual acuity measurement using Snellen's Acuity Chart and will be expressed as decimal notation
CMT(central macualr thikness ) um | 6 month
  centeral macualr thikness mesurment using using optical chorent tomgraphgy
mf-ERG amplituide nV/deg2 | 6 month
  multifocal electroretinogram amplituide mesurement using mf-ERG machine

CONTACTS AND LOCATIONS:
Locations (1):
- New Vally University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hassan A, Abdel-Radi M, Aly MOM, Alattar S. Correlation between multifocal electroretinogram and optical coherence tomography findings with visual acuity after vitrectomy surgery for retinal detachment: an observational study. Int J Retina Vitreous. 2024 Jan 23;10(1):10. doi: 10.1186/s40942-024-00527-7. PMID 38263142